CLINICAL TRIAL: NCT04354441
Title: Randomized Trial Evaluating Effect of Outpatient Hydroxychloroquine on Reducing Hospital Admissions in Pregnant Women With SARS-CoV-2 Infection: HyPreC Trial
Brief Title: Effect of Hydroxychloroquine in COVID-19 Positive Pregnant Women
Acronym: HyPreC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not started
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Haim Abenhaim, Obstetrician & gynecologist; Director of Perinatal Research, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1, March 30, 2020
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; SARS-CoV-2; Pregnant Women; Hydroxychloroquine
Keywords: COVID-19; SARS-CoV-2; Pregnancy; hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to receive either the study medication (hydroxychloroquine) or an identical-looking placebo. Randomization will be in blocks of 4-6, stratified by province.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydroxychloroquine (Experimental): 10-day course of hydroxychloroquine 200 mg tablet twice a day. To be taken orally.
  Interventions: Drug: hydroxychloroquine sulfate 200 MG
- Placebo (Placebo Comparator): An identical appearing placebo. To be taken orally twice a day for 10-days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: hydroxychloroquine sulfate 200 MG — Hydroxychloroquine sulfate (Plaquenil) 2MG will be taken twice a day for 10 days. Participants will be couriered the medication upon giving consent and will start taking the medication immediately.
  Arms: hydroxychloroquine
Drug: Placebo oral tablet — Placebo that is identical in appearance to the study medication will be taken twice a day for 10 days. It will be couriered to participants upon giving consent. They will start taking the medication immediately.
  Arms: Placebo

SUMMARY:
COVID-19 was declared a pandemic on March 11th. Efforts to save lives are essential as we will face increasing morbidity with rising demands on health care resources. Since pregnant women with COVID-19 have systematically been excluded from drug trials, potential treatment options for these high-risk individuals remain untested. The aim of our trial is to determine whether hydroxychloroquine given to COVID-19 positive pregnant women can reduce COVID-19-related hospital admissions, thereby allowing women to stay at home while limiting utilization of hospital resources and resulting exposure of health care providers.

DETAILED DESCRIPTION:
Due to physiologic and immune changes, pregnant women are at high risk of severe complications and mortality from COVID-19 infections. Despite this, epidemiologic data on SARS-CoV-2 infection in pregnancy is currently limited to small case-series describing a clinical course ranging from mild to critical illness requiring extracorporeal membrane oxygenation. Chloroquine and hydroxychloroquine (HCQ) have demonstrated activity against SARS-coronaviruses in laboratory studies and are being tested in COVID-19 positive patients. HCQ appears more promising than chloroquine due to its greater effectiveness against SARS-CoV-2 in vitro and better safety profile. To date, pregnant women have been systematically excluded from trials conducted in the general outpatient population. Thus, we will carry out a randomized, placebo-controlled, double blinded trial of HCQ (considered safe in pregnancy in pregnant women with early COVID-19 infection across Canada to evaluate its effect in reducing COVID-19-related hospitalizations. This outpatient intervention is of paramount importance as its goal is to avoid overloading emergency rooms, obstetric triage, inpatient wards and critical care units. Upon completion of 6-month, our results can be directly applied to clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Women with a self-reported live pregnancy >14 weeks
* Presently in the outpatient setting (i.e. not admitted to the hospital)
* Tested positive for COVID-19 within last 7 days
* Must be living in Canada

Exclusion Criteria:

* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Known cardiac disease (or under investigation)
* Currently taking medication contraindicated as per Health Canada list for hydroxychloroquine
* Known retinopathy
* Known hypersensitivity to 4-aminoquinoline compounds
* Already taking hydroxychloroquine
* Unwilling to answer follow-up questionnaires
* Currently in labor
* Inpatient women at time of COVID-19 diagnosis.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
COVID-19-related hospital admissions | Hospital Admission at any point from study enrollment to delivery
  COVID-19-related hospital admissions will be reported by the participants throughout pregnancy until delivery.

SECONDARY OUTCOMES:
Symptoms related to COVID-19 infection | Participants will be contacted at day 3, 7, and 10 post-randomization, and every 2 weeks up to to delivery
  Measurement of reported symptoms using a validated questionnaire on Day 3, 7, 10, and every 2 weeks. The FLU-PRO Questionnaire instructs respondents to rate the severity of 37 influenza symptoms over the past 24 hours, including those related to the nose, throat, eye, chest, head, stomach, fatigue, and body aches/pains. For 32 of 37 items, respondents rated the severity of each symptom on 5-point Likert-type scales from 0 ("Not at all), 1 ("A little bit"), 2 ("Somewhat"), 3 ("Quite a bit"), to 4 ("Very much"). For the five remaining items, severity is expressed as frequency of occurrence: vomiting or diarrhea (0 times, 1 time, 2 times, 3 times, or 4 or more times), and sneezing, coughing, and coughed up mucus or phlegm on a scale from 0 ("Never") to 4 ("Always"), with higher scores indicating more severe symptoms.
Adverse Events | Participants will be contacted at day 3, 7, and 10 post-randomization, and every 2 weeks up to to delivery
  Side effects related to hydroxychloqoruine
Maternal outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their labor and delivery.
  Type of delivery (elective non-urgent cesarean, elective urgent cesarean section, non-elective cesarean within labor, instrumental vaginal, spontaneous vaginal)
Maternal outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their labor and delivery.
  If had cesarean delivery, indication for cesarean section
Maternal outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their labor and delivery.
  Miscarriage or stillbirth (Yes/No)
Maternal outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their labor and delivery.
  Labor induction or augmentation (Yes/No) and indication
Maternal outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their labor and delivery.
  Epidural use (Yes/No)
Newborn outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their baby.
  Gestational age at delivery (weeks)
Newborn outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their baby.
  Sex (female/male)
Newborn outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their baby.
  Birth weight (kg)
  Birth weight (kg)
Newborn outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their baby.
  Need for resuscitation (Yes/No)
Newborn outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their baby.
  NICU admission (Yes/No)
Newborn outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their baby.
  Medical conditions (jaundice, IVH, RDS, pneumothorax, PDA, NEC)
Newborn outcomes | Participants will be contacted within 2 weeks after delivery to obtain information about their baby.
  Current disposition of baby (home or hospital)

REFERENCES:
- [Background] Lapinsky SE. Management of Acute Respiratory Failure in Pregnancy. Semin Respir Crit Care Med. 2017 Apr;38(2):201-207. doi: 10.1055/s-0037-1600909. Epub 2017 May 22. PMID 28561251
- [Background] Callaghan WM, Creanga AA, Jamieson DJ. Pregnancy-Related Mortality Resulting From Influenza in the United States During the 2009-2010 Pandemic. Obstet Gynecol. 2015 Sep;126(3):486-490. doi: 10.1097/AOG.0000000000000996. PMID 26244541
- [Background] Mor G, Cardenas I. The immune system in pregnancy: a unique complexity. Am J Reprod Immunol. 2010 Jun;63(6):425-33. doi: 10.1111/j.1600-0897.2010.00836.x. Epub 2010 Mar 29. PMID 20367629
- [Background] Chen H, Guo J, Wang C, Luo F, Yu X, Zhang W, Li J, Zhao D, Xu D, Gong Q, Liao J, Yang H, Hou W, Zhang Y. Clinical characteristics and intrauterine vertical transmission potential of COVID-19 infection in nine pregnant women: a retrospective review of medical records. Lancet. 2020 Mar 7;395(10226):809-815. doi: 10.1016/S0140-6736(20)30360-3. Epub 2020 Feb 12. PMID 32151335
- [Background] Liu Y, Chen H, Tang K, Guo Y. Withdrawn: Clinical manifestations and outcome of SARS-CoV-2 infection during pregnancy. J Infect. 2020 Mar 5:S0163-4453(20)30109-2. doi: 10.1016/j.jinf.2020.02.028. Online ahead of print. PMID 32145216
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Andreoli L, Bertsias GK, Agmon-Levin N, Brown S, Cervera R, Costedoat-Chalumeau N, Doria A, Fischer-Betz R, Forger F, Moraes-Fontes MF, Khamashta M, King J, Lojacono A, Marchiori F, Meroni PL, Mosca M, Motta M, Ostensen M, Pamfil C, Raio L, Schneider M, Svenungsson E, Tektonidou M, Yavuz S, Boumpas D, Tincani A. EULAR recommendations for women's health and the management of family planning, assisted reproduction, pregnancy and menopause in patients with systemic lupus erythematosus and/or antiphospholipid syndrome. Ann Rheum Dis. 2017 Mar;76(3):476-485. doi: 10.1136/annrheumdis-2016-209770. Epub 2016 Jul 25. PMID 27457513
- [Background] Izmirly PM, Costedoat-Chalumeau N, Pisoni CN, Khamashta MA, Kim MY, Saxena A, Friedman D, Llanos C, Piette JC, Buyon JP. Maternal use of hydroxychloroquine is associated with a reduced risk of recurrent anti-SSA/Ro-antibody-associated cardiac manifestations of neonatal lupus. Circulation. 2012 Jul 3;126(1):76-82. doi: 10.1161/CIRCULATIONAHA.111.089268. Epub 2012 May 24. PMID 22626746
- [Background] Costedoat-Chalumeau N, Amoura Z, Duhaut P, Huong DL, Sebbough D, Wechsler B, Vauthier D, Denjoy I, Lupoglazoff JM, Piette JC. Safety of hydroxychloroquine in pregnant patients with connective tissue diseases: a study of one hundred thirty-three cases compared with a control group. Arthritis Rheum. 2003 Nov;48(11):3207-11. doi: 10.1002/art.11304. PMID 14613284
- [Background] Costedoat-Chalumeau N, Amoura Z, Huong DL, Lechat P, Piette JC. Safety of hydroxychloroquine in pregnant patients with connective tissue diseases. Review of the literature. Autoimmun Rev. 2005 Feb;4(2):111-5. doi: 10.1016/j.autrev.2004.11.009. Epub 2004 Dec 14. PMID 15722258